CLINICAL TRIAL: NCT01205035
Title: High-Dose Lucentis (Ranibizumab 2.0mg) for the Treatment of Nonproliferative Idiopathic Parafoveal Telangiectasia [HD-LIPT]
Brief Title: High-Dose Lucentis (Ranibizumab 2.0mg) for the Treatment of Nonproliferative Idiopathic Parafoveal Telangiectasia
Acronym: HD-LIPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eye Center of Northern Colorado, P.C. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Arthur Korotkin, M.D., M.D., Eye Center of Northern Colorado, P.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4875s
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Retinal Diseases; Telangiectasis
Keywords: Idiopathic Parafoveal Telangiectasia; Macular Telangiectasia; Macula Lutea/pathology; Retinal Diseases/pathology; Retinal Pigments/metabolism; Telangiectasis/metabolism; Telangiectasis/pathology
MeSH Terms: conditions — Retinal Diseases; Telangiectasis | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (No Intervention): Observation; No treatment given
- Intravitreal ranibizumab 2.0mg (Experimental): Initial dose 2.0mg switched to 1.0mg at near conclusion of study.
  Interventions: Drug: ranibizumab 2.0mg

INTERVENTIONS:
Drug: ranibizumab 2.0mg — Baseline monthly intravitreal injection of ranibizumab 2.0mg for 3 months followed by possible monthly injections up to 9 additional injections
  Other Names: Lucentis
  Arms: Intravitreal ranibizumab 2.0mg

SUMMARY:
Idiopathic Parafoveal Telangiectasia (IPT) [also known as Idiopathic Perifoveal Telangiectasia, Idiopathic Juxtafoveal Telangiectasia (IJT, JFT) and Macular Telangiectasia (MacTel)] is a disorder of unknown etiology. IPT is classified as Group 2A in the Gass classification of macular telangiectasias (Reference 1,5) - a bilateral, but not always symmetric disorder. It is characterized in its early stages by dilation and loss of parafoveal capillaries accompanied by angiographic leakage, "right angle" venules, central and parafoveal intraretinal cysts.

DETAILED DESCRIPTION:
DESCRIPTION OF THE STUDY

This is an open-label, Phase I/II study of intravitreally administered ranibizumab in subjects with nonproliferative Idiopathic Parafoveal Telangiectasia (IPT).

Consented, enrolled subjects will be randomized into two groups: observation and treatment. The observation group will be monitored monthly while the treatment group will receive three open-label intravitreal injections of 1.0 mg ranibizumab administered every 30 days for 3 months and then as needed monthly, based on defined criteria. NOTE: The original protocol had the treatment group dosed at 2.0 mg/0.05mL. However, the 2.0mg dose will become unavailable beginning January 31, 2012. Therefore, the protocol amendment submitted in December 2011 changed the 2.0mg arm to a 1.0mg/ 0.10mL arm. Please note that three patients were already treated with 2.0mg before the amendment was submitted, so they will be switched to 1.0mg if they have not completed the study when the 2.0 dose is no longer available in January 2012.

Protocol: FVF4875s Final 6/P

29MAR2010

3.2

RATIONALE FOR STUDY DESIGN

As IPT is a chronically progressive condition, the purpose of this study is to see if high-dose ranibizumab can slow or stop the leakage and growth of existing, dilated, macular vessels in cases where no co-existing neovascularization exists as defined by fluorescein angiography and Ocular Coherence Tomography (OCT). Other outcomes include stabilization of visual acuity compared to observation group (defined by best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) measurements), and changes in ultrastructural features, as defined by OCT,

3.3

OUTCOME MEASURES

3.3.1 Primary Outcome Measures

To compare the change in visual acuity from baseline to one year in patients with nonproliferative IPT who are either treated with high-dose (1.0mg) ranibizumab or observed.

3.3.2 Secondary Outcome Measures

i. To compare the change in visual acuity from baseline to 6 months and 9 months in patients with nonproliferative IPT who are either treated with high- dose (1.0mg) ranibizumab or observed.

ii. To assess OCT changes in standard Central Subfield Thickness (CST) from baseline to 6 months, 9 months and 12 months.

iii. To assess safety of administering 1.0mg ranibizumab (Lucentis) in patients with nonproliferative IPT at 6 months, 9 months and 12 months.

iv. To assess changes in angiographic leakage from baseline at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Presence of nonproliferative IPT confirmed by fluorescein angiography and spectral-domain OCT
* Age greater than 18
* Vision equal to or worse than 20/25 and better than or equal to 20/400 by ETDRS chart, without co-existing choroidal neovascularization.
* Physical ability and reasonable expectation to maintain all follow-up appointments.

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous ophthalmologic investigation or trial
* Any patient with proliferative diabetic retinopathy, diabetic macular edema, uveitis, history of ocular trauma, severe glaucoma, neovascular age-related macular degeneration
* Duration of previous treatment of IPT that exceeds two years.
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either:
* Require medical or surgical intervention during the 12-month study period to prevent or treat visual loss that might result from that condition, or
* If allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of Best Corrected Visual Acuity (BCVA) over the study period
* Prior/Concomitant Treatment:
* Previous steroids (oral) within 30 days preceding Day 0
* Previous participation in any studies of investigational drugs within 30 days preceding Day 0 (excluding vitamins and minerals)
* Prior participation in a Genentech ranibizumab clinical trial within 60 days.
* History of receiving intravitreal injections of ranibizumab, bevacizumab, pegaptanib, or any other intravitreal medication within 60 days of first injection. History of receiving intravitreal or subtenons triamcinolone within 90 days of first injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Korotkin, M.D., Principal Investigator — Eye Center of Northern Colorado
Locations (1):
- Eye Center of Northern Colorado, Fort Collins, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg
Started | 3 | 3
Completed | 1 | 3
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 68 [52 to 76] | 65 [52 to 76] | 66.5 [52 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Change From Baseline to Month 12 of the Study
Time Frame: Baseline to 12 months
Measure: Mean (Full Range); unit: LogMAR Unit
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg
Number analyzed (Participants) | 1 | 3
LogMAR Unit | 0.1 [0.1 to 0.1] | -0.05 [-0.12 to 0]

2. Secondary Outcome: Change in Visual Acuity From Baseline to Month 6 and From Baseline to 9 Months
Time Frame: Baseline to 6 months and baseline to 9 months
Measure: Mean (Full Range); unit: LogMAR Unit
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg
Number analyzed (Participants) | 1 | 3
LogMAR Unit
  Baseline to 6 month | 0.04 [0.04 to 0.04] | -0.10 [-0.2 to -0.02]
  Baseline to 9 month | 0.02 [0.02 to 0.02] | -0.12 [-0.14 to -0.08]

3. Secondary Outcome: Change in Standard Central Subfield Thickness (CST) as Measured by OCT From Baseline to 6, 9, and 12 Months
Description: A large decrease in CST thickness may be indicative of a worse clinical outcome. These measurements are done to ensure safety of the participants.
Time Frame: Baseline to 6, 9, and 12 months
Measure: Mean (Full Range); unit: Micrometer
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg
Number analyzed (Participants) | 1 | 3
Micrometer
  Baseline to 6 month | -20 [-20 to -20] | 7 [-2 to 20]
  Baseline to 9 month | -16 [-16 to -16] | -6 [-17 to 12]
  Baseline to 12 month | -11 [-11 to -11] | -4 [-14 to 2]

4. Secondary Outcome: Number of Adverse Events Associated to the Administration of Ranibizumab 2.0mg
Time Frame: Baseline to 6 month, baseline to 9 month and baseline to 12 months
Measure: Number; unit: Number of Adverse Events
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg
Number analyzed (Participants) | 1 | 3
Number of Adverse Events
  Baseline to 6 month | 0 | 0
  Baseline to 9 month | 0 | 0
  Baseline to 12 month | 0 | 0

5. Secondary Outcome: Angiographic Leakage From Baseline to Month 6 and 12
Description: Angiography was taken via fluorescein angiography. Any increases of angiographic leakage was counted between baseline and month 6. Also any decreases of angiographic leakage was counted between baseline and 6 month. The same was done between baseline and 12 month.
  Any increase of angiographic leakage was counted as a +1. Likewise, any decrease of angiographic leakage was counted as a -1. The sum was calculated based on the number of participants in each arm and the total shown in the outcome. For example: if across the three injected participants for their 6 month visit, two of them showed an increase of angiographic leakage and one showed a decrease, then the outcome would be, (+1) + (+1) + (-1)= +1. Likewise, if the same three participant's 12 month visit showed two with a decrease in leakage and one with no changes in leakage, the outcome would be, (-1) + (-1) + (0)= -2
Time Frame: Baseline to 6 and baseline to 12 months
Measure: Number; unit: Sum of increases (+1) and decreases (-1)
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg
Number analyzed (Participants) | 1 | 3
Sum of increases (+1) and decreases (-1)
  Baseline to 6 month | 0 | 1
  Baseline to 12 month | 0 | -2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Observation | Intravitreal Ranibizumab 2.0mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation (N=3) | Intravitreal Ranibizumab 2.0mg (N=3)
Elevated Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Cold (Immune system disorders) | 1 (1) | 0 (0)
Food Poisoning (General disorders) | 1 (1) | 0 (0)
Diabetes (Endocrine disorders) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stiff Neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No